CLINICAL TRIAL: NCT03133065
Title: Early Treatment of Recurrent HCV- Infection Post Liver Transplantation in the Era of DAAs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Iman Fawzy Montasser, Clinical professor, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCV treatment
Record Dates: First submitted 2017-04-23; First posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: treatment after 6 months post transplantation (Active Comparator): 53 patients received Sofosbuvir+ribavirin standard of care for treatment of HCV post liver transplantation for 6 months
  Interventions: Drug: treatment of HCV with oral direct acting antiviral therapy
- Group 2: early treatment afer 3 months post transplantation (Active Comparator): 36 patients received other DAAs regiment for treatment of HCV post liver transplantation for 3- 6 months
  Interventions: Drug: treatment of HCV with oral direct acting antiviral therapy

INTERVENTIONS:
Drug: treatment of HCV with oral direct acting antiviral therapy — A total number of 89 patients transplanted for HCV genotype 4 related end stage liver disease Were included in this study 53 PATIENTS were treated after 6 months of transplantation with sofosbuvir 400mg and weight based ribavirin for 24 weeks. 7 patients were treated with sofosbuvir 400mg + simeprevir 150 mg + weight based ribavirin for 12 weeks after 6 months post transplant. In September 2015, we started to adopt early treatment strategy for all recipients after the first 3months post- transplant. 26 recipients were treated with sofosbuvir 400mg+Daclatasvir 60mg ± weight based ribavirin for 12 weeks or 24 weeks. 2 recipient are treated with sofosbuvir 400mg + ledipasvir 90mg for 24 weeks and one recipient is treated with fixed-dose combination of ombitasvir (12.5 mg), paritaprevir (75 mg) and ritonavir (50 mg) + weight based ribavirin due to having persistent renal impairment post transplantation.

SUMMARY:
The study aimed to present our experience in treating recurrent HCV genotype 4 infection post living donor liver transplantation (LDLT) since introduction of the second generation direct acting antiviral drugs (DAAs) in Egypt.

DETAILED DESCRIPTION:
This was a cohort study conducted in patients who had undergone LDLT for HCV related disease from 2014 to 2016 at in Ain Shams Center for Organ Transplantation (ASCOT) .The hypothesis early initiation of DAAs( after 12 weeks of the operation ) is effective and safe strategy in transplant recipients following LDLT. Patients who take the sofosbuvir and ribavirin after 6 months after transplantation were compared with those who take early treatment after 3 months of transplantation with sofosbuvir and daclatsvir+/- ribavirin..Patients were on regular follow up visits monthly to assess the clinical condition, any side effects, laboratory tests including complete blood picture, liver functions , renal functions and trough level of immunosuppressant drugs.

ELIGIBILITY:
Inclusion Criteria:

* All transplanted patients for HCV related disease in the period from 2014 to 2016

Exclusion Criteria:

* Patients transplanted for other causes rather than HCv
* Patients with HBV and HCV co infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Virologic response at 12 weeks after completion of therapy | 3 months
  Assessment of virologic response after 3 months

IPD SHARING:
Plan to Share IPD: Undecided